CLINICAL TRIAL: NCT02489266
Title: A Phase I Trial for the Evaluation of the In Vivo Persistence of Adoptively-transferred Tumor-Infiltrating Lymphocytes Cultured With a Pharmacologic Inhibitor of AKT in Patients With Metastatic Melanoma
Brief Title: In Vivo Persistence of Adoptively-Transferred TIL Cultured With Akti in People With Metastatic Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150153; 15-C-0153
Record Dates: First submitted 2015-07-02; First posted 2015-07-03 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2016-06-29

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma; Immunotherapy
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine; aldesleukin

ARMS (1):
- Arm 1 (Experimental): Patients will receive cyclophosphamide and fludarabine followed by infusion of the AKTi-treated TIL, followed by high dose aldesleukin.
  Interventions: Biological: AKTi-treated TIL; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin

INTERVENTIONS:
Biological: AKTi-treated TIL — On day 0, cells will be infused intravenously (IV) over 20-30 minutes (between 1 and 4 days after the last dose of fludarabine).
Drug: Cyclophosphamide — Patients will receive Cyclophosphamide 60 mg/kg/day x 2 days.
Drug: Fludarabine — Patients will receive Fludarabine 25 mg/m2/day for 5 days.
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).

SUMMARY:
Background:

- One cancer therapy involves taking white blood cells from a person, changing them in a lab, and then giving the cells back to the person. These cells are called tumor infiltrating lymphocytes (TIL). Researchers want to grow some of the TIL cells with the drug Akti to see if they live longer than those grown without it.

Objectives:

- To see if TIL cells grown with Akti live longer than those grown without it.

Eligibility:

- Adults 18 70 with metastatic melanoma

Design:

* Participants will:
* Be screened with tests including scans, x-rays, heart and lung tests, blood and urine tests, and a <TAB>possible colonoscopy.
* Have tumor surgery or biopsy.
* Have a large catheter inserted into a vein in the upper chest.
* Receive leukapheresis for 4 5 hours. Blood is removed through a needle in an arm. White blood cells <TAB>are removed. The rest of the blood is returned by needle in the other arm.
* The cells will be changed in a laboratory.
* Participants will check into the hospital and:
* For 5 days, get 1 2 chemotherapy drugs by catheter.
* For 1 3 days, get the changed cells by catheter.
* For several days, get 2 drugs to stimulate cells, one by injection, the other by catheter.
* For 7 12 days, recover in the hospital.
* After treatment, participants will:
* Take an antibiotic and antiviral for at least 6 months.
* Return to NIH for several 2-day visits for a few years. At each visit, participants will have lab tests, imaging studies, and a physical exam. At some visits, they may have leukapheresis or blood tests.

DETAILED DESCRIPTION:
Background:

* Adoptive cellular immunotherapy (ACT) using autologous tumor-infiltrating lymphocytes (TIL) can mediate regression of bulky metastatic melanoma when administered with high-dose aldesleukin (IL-2) following a non-myeloablative lymphodepleting chemotherapy preparative regimen consisting of cyclophosphamide and fludarabine.
* Regression of tumor in mouse models and humans strongly correlates with anti-tumor T cells that exhibit features of immunologic memory and have a capacity to persist for long periods after adoptive-transfer into tumor-bearing hosts.
* In our preclinical work with TIL, we have identified a pharmacologic inhibitor of AKT that promotes features of immunologic memory in TIL (as evidenced by transcriptomic, proteomic, metabolomic, and functional assays described in the Background section). Consistently, AKT inhibition of human TIL significantly enhances persistence after adoptive-transfer into an immunodeficient mouse model.
* We therefore aim to evaluate whether pharmacologic inhibition of AKT in TIL may enhance persistence after adoptive-transfer into patients with advanced melanoma.

Objectives:

* Primary objective:

  * To determine whether ACT using TIL cultured in a pharmacologic inhibitor of AKT (during ex vivo expansion) results in enhanced in vivo persistence of TIL after adoptive transfer into autologous patients with advanced melanoma.
* Secondary objectives:

  * Determine the toxicity profile of this treatment regimen.
  * Determine whether ACT using a combination of AKTi-treated and conventional TIL can mediate tumor regression by RECIST (Response Evaluation Criteria in Solid Tumors) guidelines in patients with advanced melanoma.

Eligibility:

* Age greater than or equal to 18 and less than or equal to 70 years
* Evaluable metastatic melanoma
* Metastatic melanoma lesion suitable for surgical resection for the preparation of TIL
* No contraindications to high-dose aldesleukin administration
* No concurrent major medical illnesses or any form of immunodeficiency

Design:

* Patients with metastatic melanoma will undergo ACT in conventional manner, with the exception that half of tumor fragments from which TIL are isolated will be cultured in the presence of a pharmacologic AKT inhibitor. Prior to infusion of TIL, the AKT inhibitor (hereafter AKTi) will be washed from the therapeutic TIL product and will not be systemically administered. Each patient will receive a 1:1 mixture of conventional TIL and AKTi-treated TIL. To evaluate persistence of AKTi-treated and conventional TIL after adoptive co-transfer, we will perform high-throughput deep sequencing of the TCR V-beta CDR3 region of TIL from the infusion-bag and from peripheral blood when sufficient lymphocyte reconstitution (>200 lymphocytes/microliter) has occurred and approximately 4-6 weeks after infusion.
* Up to 20 patients may be enrolled over 20-24 months.

ELIGIBILITY:
* INCLUSION CRITERIA
* Measurable metastatic melanoma with at least one lesion that is resectable for TIL generation, plus one other lesion that can be measured.
* Confirmation of diagnosis of metastatic melanoma by the Laboratory of Pathology of NCI.
* Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
* Prior therapy with at least one first line standard therapy including check point inhibitors such as pembrolizumab, nivolumab, or ipilimumab.

  * Note: Six weeks must have elapsed from the time of any of these prior antibody therapies that could affect an anti-cancer immune response, at the time the patient receives the preparative regimen to allow antibody levels to decline.
  * Note: Patients who have previously received ipilimumab and have documented GI toxicity must have a normal colonoscopy with normal colonic biopsies.
* Greater than or equal to 18 years of age and less than or equal to 70 years of age.
* Willing to sign a durable power of attorney.
* Able to understand and sign the Informed Consent Document
* Clinical performance status of ECOG 0 or 1.
* Life expectancy of greater than three months.
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
* Serology:

  * Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
* Hematology:

  * Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim
  * WBC greater than or equal to 3000/mm^3
  * Platelet count greater than or equal to 100,000/mm^3
  * Hemoglobin > 8.0 g/dl
* Chemistry:

  * Serum ALT/AST less than or equal to 2.5 times the upper limit of normal
  * Serum Creatinine less than or equal to 1.6 mg/dl
  * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert s Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients must have progressive disease after prior treatment.

  * Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.
* Six weeks must have elapsed from the time of any antibody therapy that could affect an anti cancer immune response, including anti-CTLA4 antibody therapy, at the time the patient receives the preparative regimen to allow antibody levels to decline.

  * Note: Patients who have previously received ipilimumab and have documented GI toxicity must have a colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA

* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Active systemic infections (for e.g.: requiring anti-infective treatment), coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Concurrent systemic steroid therapy.
* History of severe immediate hypersensitivity reaction to cyclophosphamide or fludarabine.
* History of coronary revascularization or ischemic symptoms.
* Documented LVEF of less than or equal to 45%, testing is required in patients with:

  * Age greater than or equal to 60 years old
  * Clinically significant atrial and or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06-24; Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

PRIMARY OUTCOMES:
Determine whether ACT using TIL cultured in a pharmacologic inhibitor of AktKT (during ex vivo expansion) results in enhanced in vivo persistence of TIL after adoptive transfer into autologous patients with advanced melanoma. | 4 years

SECONDARY OUTCOMES:
Determine whether ACT using a combination of conventional and AKTi-treated TIL can mediate tumor regression by RECIST guidelines in patients with advanced melanoma | 4 years
Determine the toxicity profile of this treatment regimen. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Rosenberg SA, Yang JC, Sherry RM, Kammula US, Hughes MS, Phan GQ, Citrin DE, Restifo NP, Robbins PF, Wunderlich JR, Morton KE, Laurencot CM, Steinberg SM, White DE, Dudley ME. Durable complete responses in heavily pretreated patients with metastatic melanoma using T-cell transfer immunotherapy. Clin Cancer Res. 2011 Jul 1;17(13):4550-7. doi: 10.1158/1078-0432.CCR-11-0116. Epub 2011 Apr 15. PMID 21498393
- [Background] Robbins PF, Morgan RA, Feldman SA, Yang JC, Sherry RM, Dudley ME, Wunderlich JR, Nahvi AV, Helman LJ, Mackall CL, Kammula US, Hughes MS, Restifo NP, Raffeld M, Lee CC, Levy CL, Li YF, El-Gamil M, Schwarz SL, Laurencot C, Rosenberg SA. Tumor regression in patients with metastatic synovial cell sarcoma and melanoma using genetically engineered lymphocytes reactive with NY-ESO-1. J Clin Oncol. 2011 Mar 1;29(7):917-24. doi: 10.1200/JCO.2010.32.2537. Epub 2011 Jan 31. PMID 21282551
- [Background] Tran E, Turcotte S, Gros A, Robbins PF, Lu YC, Dudley ME, Wunderlich JR, Somerville RP, Hogan K, Hinrichs CS, Parkhurst MR, Yang JC, Rosenberg SA. Cancer immunotherapy based on mutation-specific CD4+ T cells in a patient with epithelial cancer. Science. 2014 May 9;344(6184):641-5. doi: 10.1126/science.1251102. PMID 24812403